Document: TDOC-0056910 Version: 2.0; Most-Recent; Effective; CURRENT

Status: Effective 

Title

# Clinical Evaluation of a Daily Wear Monthly Replacement Silicone Hydrogel Lens

Protocol Number: CLY935-C010 / NCT04178720

Development Stage of

Development

Project:

Sponsor Name and Alcon Research, LLC and its affiliates ("Alcon")

Address: 6201 South Freeway

Fort Worth, Texas 76134-2099

Test Product: LID018869

Property of Alcon
Confidential
May not be used, divulged, published, or otherwise disclosed without the consent of
Alcon


Status: Effective 

#### Investigator Agreement:

• I have read the clinical study described herein, recognize its confidentiality, and agree to conduct the described trial in compliance with Good Clinical Practice (GCP), the ethical principles contained within the Declaration of Helsinki, this protocol, all applicable regulatory authority regulations, and conditions of approval imposed by the reviewing IRB or regulatory authority.

- I will supervise all testing of the device involving human subjects and ensure that the requirements relating to obtaining informed consent and IRB review and approval are met in accordance with applicable local and governmental regulations.
- I have read and understand the appropriate use of the investigational product(s) as described in the protocol, current Investigator's Brochure, product information, or other sources provided by the Sponsor.
- I understand the potential risks and side effects of the investigational product(s).
- I agree to maintain adequate and accurate records in accordance with government regulations and to make those records available for inspection.
- I agree to comply with all other requirements regarding the obligations of clinical Investigators and all other pertinent requirements of the Sponsor and government agencies.
- I agree to ensure that all associates, colleagues, and employees assisting in the conduct of the study are informed of their obligations in meeting the above commitments.

| Have you ever been | disqualified as an Investigator b | y any Regulatory Authority? |
|---|---|---|
| □ No □Yes | | |
| Have you ever been | involved in a study or other rese | earch that was terminated? |
| □ No □Yes | | |
| If yes, please explain | n here: | |
| L | | |
| Principal Investigator: | | |
| | Signature | Date |
| Name and professional position: | | |
| Address: | | |


Status: Effective 

Effective Date: 08-Nov-2019

# **Table of Contents**

| Cl | inical Eva | lluation of a Daily Wear Monthly Replacement Silicone Hydrogel Lens | 1 |
|---|---|---|---|
| Та | ble of Co | ntents | |
| Li | st of Table | es | 4 |
| Li | st of Figu | res | |
| 1 | _ | ARY OF TERMS | |
| 2 | LIST OF | F ACRONYMS AND ABBREVIATIONS | 1 |
| 3 | PROTO | COL SUMMARY | 13 |
| 4 | | COL AMENDMENTS | |
| | 4.1 | Amendments | |
| 5 | | DUCTION | |
| | 5.1 | Rationale and Background | |
| | 5.2 | Purpose of the Study | |
| | 5.3 | Risks and Benefits | |
| 6 | STUDY | OBJECTIVES | 25 |
| | 6.1 | Primary Objective(s) | 25 |
| | 6.2 | Secondary Objective(s) | 25 |
| | 6.4 | Safety Objective(s) | 25 |
| 7 | INVEST | TIGATIONAL PLAN | 25 |
| | 7.1 | Study Design | 25 |
| | 7.2 | Rationale for Study Design | 27 |
| | 7.3 | Rationale for Duration of Treatment/Follow-Up | 27 |
| | 7.4 | Rationale for Choice of Control Product | 27 |
| | 7.5 | Data Monitoring Committee | 27 |
| 8 | STUDY | POPULATION | 27 |
| | 8.1 | Inclusion Criteria | 28 |
| | 8.2 | Exclusion Criteria | 29 |
| | 8.3 | Rescreening of Subjects | 30 |
| 9 | TREAT | MENTS ADMINISTERED | 30 |
| | 9.1 | Investigational Product(s) | 30 |

| Page 4 of 66 | | usiness Use Only Protocol - Clinical Effective Date: 08-Nov | v-2019 |
|---|---|---|---|
| 9.3 Treatment Masking | | | <b>4</b> of <b>6</b> 0 |
| 9.4 Treatment Masking | 9.2 | Other Medical Device or Medication Specified for Use During the Study. | 35 |
| 9.4 Treatment Masking | 9.3 | Treatment Assignment/Randomization | 36 |
| 9.6 Changes to Concomitant Medications, Treatments/Procedures 35 10 STUDY PROCEDURES AND ASSESSMENTS 35 10.1 Informed Consent and Screening 40 10.2 Description of Study Procedures and Assessments 41 10.2.1 Demographics 41 10.2.2 Medical History 41 10.2.3 Investigational Product Compliance 41 10.2.4 Adverse Event Collection: Safety Assessment 41 10.2.5 Slit-Lamp Biomicroscopy: Safety Assessment 41 10.2.6 Device Deficiencies: Safety Assessment 41 10.2.7 Visual Acuity: Effectiveness Assessment 42 10.3 Additional Study Assessments 42 10.4 Unscheduled Visits 42 10.5 Discontinued Subjects 43 10.5 Discontinued Subjects 43 10.5 Discontinuations 43 10.5 Discontinuations 43 10.5 Schedule of Procedures and Assessments for Subjects Discontinued from Investigational Product 44 10.6 Clinical Study Termination 44 | 9.4 | | |
| 9.6 Changes to Concomitant Medications, Treatments/Procedures 35 10 STUDY PROCEDURES AND ASSESSMENTS 35 10.1 Informed Consent and Screening 40 10.2 Description of Study Procedures and Assessments 41 10.2.1 Demographics 41 10.2.2 Medical History 41 10.2.3 Investigational Product Compliance 41 10.2.4 Adverse Event Collection: Safety Assessment 41 10.2.5 Slit-Lamp Biomicroscopy: Safety Assessment 41 10.2.6 Device Deficiencies: Safety Assessment 41 10.2.7 Visual Acuity: Effectiveness Assessment 42 10.3 Additional Study Assessments 42 10.4 Unscheduled Visits 42 10.5 Discontinued Subjects 43 10.5 Discontinued Subjects 43 10.5 Discontinuations 43 10.5 Discontinuations 43 10.5 Schedule of Procedures and Assessments for Subjects Discontinued from Investigational Product 44 10.6 Clinical Study Termination 44 | 9.5 | Accountability Procedures | 38 |
| 10 STUDY PROCEDURES AND ASSESSMENTS 36 10.1 Informed Consent and Screening 40 10.2 Description of Study Procedures and Assessments 41 10.2.1 Demographics 41 10.2.2 Medical History 41 10.2.3 Investigational Product Compliance 41 10.2.4 Adverse Event Collection: Safety Assessment 41 10.2.5 Slit-Lamp Biomicroscopy: Safety Assessment 41 10.2.6 Device Deficiencies: Safety Assessment 41 10.2.7 Visual Acuity: Effectiveness Assessment 42 10.3 Additional Study Assessments 42 10.4 Unscheduled Visits 42 10.5 Discontinued Subjects 43 10.5.1 Screen Failures 43 10.5.2 Discontinuations 43 10.5.3 Schedule of Procedures and Assessments for Subjects Discontinued from Investigational Product 44 10.6 Clinical Study Termination 44 10.6.1 Follow-up of Subjects After Study Participation Has Ended 45 11.1 General Information 45 11.2 Monitoring for AEs 45 11.3 Procedures for Recording and Reporting 48 11.4 Return Product Analysis 51 11.5 Unmasking | 9.6 | - | |
| 10.2 Description of Study Procedures and Assessments .41 10.2.1 Demographics .41 10.2.2 Medical History .41 10.2.3 Investigational Product Compliance .41 10.2.4 Adverse Event Collection: Safety Assessment .41 10.2.5 Slit-Lamp Biomicroscopy: Safety Assessment .41 10.2.6 Device Deficiencies: Safety Assessment .41 10.2.7 Visual Acuity: Effectiveness Assessment .42 10.3 Additional Study Assessments .42 10.4 Unscheduled Visits .42 10.5 Discontinued Subjects .42 10.5.1 Screen Failures .42 10.5.2 Discontinuations .43 10.5.3 Schedule of Procedures and Assessments for Subjects Discontinued from Investigational Product .44 10.6 Clinical Study Termination .44 10.6.1 Follow-up of Subjects After Study Participation Has Ended .45 11.1 General Information .45 11.2 Monitoring for AEs .48 11.3 Procedures for Recording and Reporting .48 <td>10 STUD</td> <td>-</td> <td></td> | 10 STUD | - | |
| 10.2 Description of Study Procedures and Assessments .41 10.2.1 Demographics .41 10.2.2 Medical History .41 10.2.3 Investigational Product Compliance .41 10.2.4 Adverse Event Collection: Safety Assessment .41 10.2.5 Slit-Lamp Biomicroscopy: Safety Assessment .41 10.2.6 Device Deficiencies: Safety Assessment .41 10.2.7 Visual Acuity: Effectiveness Assessment .42 10.3 Additional Study Assessments .42 10.4 Unscheduled Visits .42 10.5 Discontinued Subjects .42 10.5.1 Screen Failures .42 10.5.2 Discontinuations .43 10.5.3 Schedule of Procedures and Assessments for Subjects Discontinued from Investigational Product .44 10.6 Clinical Study Termination .44 10.6.1 Follow-up of Subjects After Study Participation Has Ended .45 11.1 General Information .45 11.2 Monitoring for AEs .48 11.3 Procedures for Recording and Reporting .48 <td>10.</td> <td>1 Informed Consent and Screening</td> <td>40</td> | 10. | 1 Informed Consent and Screening | 40 |
| 10.2.1 Demographics. .41 10.2.2 Medical History. .41 10.2.3 Investigational Product Compliance. .41 10.2.4 Adverse Event Collection: Safety Assessment .41 10.2.5 Slit-Lamp Biomicroscopy: Safety Assessment .41 10.2.6 Device Deficiencies: Safety Assessment .41 10.2.7 Visual Acuity: Effectiveness Assessment .42 10.3 Additional Study Assessments .42 10.4 Unscheduled Visits .42 10.5 Discontinued Subjects .42 10.5 Discontinuations .43 10.5.2 Discontinuations .43 10.5.3 Schedule of Procedures and Assessments for Subjects Discontinued from Investigational Product .44 10.6 Clinical Study Termination .44 10.6.1 Follow-up of Subjects After Study Participation Has Ended .45 11.1 General Information .45 11.2 Monitoring for AEs .48 11.3 Procedures for Recording and Reporting .48 11.4 Return Product Analysis .51 | 10. | - | |
| 10.2.2 Medical History 41 10.2.3 Investigational Product Compliance 41 10.2.4 Adverse Event Collection: Safety Assessment 41 10.2.5 Slit-Lamp Biomicroscopy: Safety Assessment 41 10.2.6 Device Deficiencies: Safety Assessment 41 10.2.7 Visual Acuity: Effectiveness Assessment 42 10.3 Additional Study Assessments 42 10.4 Unscheduled Visits 42 10.5 Discontinued Subjects 43 10.5.1 Screen Failures 43 10.5.2 Discontinuations 42 10.5.3 Schedule of Procedures and Assessments for Subjects Discontinued from Investigational Product 44 10.6 Clinical Study Termination 44 10.6.1 Follow-up of Subjects After Study Participation Has Ended 45 11 ADVERSE EVENTS AND DEVICE DEFICIENCIES 45 11.1 General Information 45 11.2 Monitoring for AEs 48 11.3 Procedures for Recording and Reporting 48 11.4 Return Product Analysis 51 11.5 Unmasking of the Study Treatment 51 11.6 Follow-Up of Subjects with AEs 51 11.7 Pregnancy in the Clinical Study 51 | | | |
| 10.2.3 Investigational Product Compliance | | | |
| 10.2.4 Adverse Event Collection: Safety Assessment 41 10.2.5 Slit-Lamp Biomicroscopy: Safety Assessment 41 10.2.6 Device Deficiencies: Safety Assessment 41 10.2.7 Visual Acuity: Effectiveness Assessment 42 10.3 Additional Study Assessments 42 10.4 Unscheduled Visits 42 10.5 Discontinued Subjects 43 10.5.1 Screen Failures 43 10.5.2 Discontinuations 43 10.5.2 Discontinuations 43 10.5.3 Schedule of Procedures and Assessments for Subjects Discontinued from Investigational Product 44 10.6 Clinical Study Termination 44 10.6.1 Follow-up of Subjects After Study Participation Has Ended 45 11 ADVERSE EVENTS AND DEVICE DEFICIENCIES 45 11.1 General Information 45 11.2 Monitoring for AEs 48 11.3 Procedures for Recording and Reporting 48 11.4 Return Product Analysis 51 11.5 Unmasking of the Study Treatment 51 | | ž | |
| 10.2.5 Slit-Lamp Biomicroscopy: Safety Assessment .41 10.2.6 Device Deficiencies: Safety Assessment .41 10.2.7 Visual Acuity: Effectiveness Assessment .42 10.3 Additional Study Assessments .42 10.4 Unscheduled Visits .42 10.5 Discontinued Subjects .43 10.5.1 Screen Failures .43 10.5.2 Discontinuations .43 10.5.3 Schedule of Procedures and Assessments for Subjects Discontinued from Investigational Product .44 10.6 Clinical Study Termination .44 10.6.1 Follow-up of Subjects After Study Participation Has Ended .45 11 ADVERSE EVENTS AND DEVICE DEFICIENCIES .45 11.1 General Information .45 11.2 Monitoring for AEs .45 11.3 Procedures for Recording and Reporting .48 11.4 Return Product Analysis .51 11.5 Unmasking of the Study Treatment .51 11.6 Follow-Up of Subjects with AEs .51 11.7 Pregnancy in the Clinical Study .51 | | | |
| 10.2.7 Visual Acuity: Effectiveness Assessment 42 10.3 Additional Study Assessments 42 10.4 Unscheduled Visits 42 10.5 Discontinued Subjects 43 10.5.1 Screen Failures 43 10.5.2 Discontinuations 42 10.5.3 Schedule of Procedures and Assessments for Subjects Discontinued from Investigational Product 44 10.6 Clinical Study Termination 44 10.6.1 Follow-up of Subjects After Study Participation Has Ended 45 11 ADVERSE EVENTS AND DEVICE DEFICIENCIES 45 11.1 General Information 45 11.2 Monitoring for AEs 48 11.3 Procedures for Recording and Reporting 48 11.4 Return Product Analysis 51 11.5 Unmasking of the Study Treatment 51 11.6 Follow-Up of Subjects with AEs 51 11.7 Pregnancy in the Clinical Study 51 | | | |
| 10.3 Additional Study Assessments | | 10.2.6 Device Deficiencies: Safety Assessment | 41 |
| 10.4 Unscheduled Visits 42 10.5 Discontinued Subjects 43 10.5.1 Screen Failures 43 10.5.2 Discontinuations 43 10.5.3 Schedule of Procedures and Assessments for Subjects Discontinued from Investigational Product 44 10.6 Clinical Study Termination 44 10.6.1 Follow-up of Subjects After Study Participation Has Ended 45 11 ADVERSE EVENTS AND DEVICE DEFICIENCIES 45 11.1 General Information 45 11.2 Monitoring for AEs 48 11.3 Procedures for Recording and Reporting 48 11.4 Return Product Analysis 51 11.5 Unmasking of the Study Treatment 51 11.6 Follow-Up of Subjects with AEs 51 11.7 Pregnancy in the Clinical Study 51 | | 10.2.7 Visual Acuity: Effectiveness Assessment | 42 |
| 10.5 Discontinued Subjects | 10. | 3 Additional Study Assessments | 42 |
| 10.5.1 Screen Failures | 10. | 4 Unscheduled Visits | 42 |
| 10.5.2 Discontinuations | 10. | 5 Discontinued Subjects | 43 |
| 10.5.2 Discontinuations | | 10.5.1 Screen Failures | 43 |
| from Investigational Product | | | |
| 10.6 Clinical Study Termination | | | |
| 11.1 General Information | 10. | | |
| 11.1 General Information | | 10.6.1 Follow-up of Subjects After Study Participation Has Ended | 45 |
| 11.2 Monitoring for AEs4811.3 Procedures for Recording and Reporting4811.4 Return Product Analysis5111.5 Unmasking of the Study Treatment5111.6 Follow-Up of Subjects with AEs5111.7 Pregnancy in the Clinical Study51 | 11 ADVE | | |
| 11.3 Procedures for Recording and Reporting4811.4 Return Product Analysis5111.5 Unmasking of the Study Treatment5111.6 Follow-Up of Subjects with AEs5111.7 Pregnancy in the Clinical Study51 | 11. | 1 General Information | 45 |
| 11.3 Procedures for Recording and Reporting4811.4 Return Product Analysis5111.5 Unmasking of the Study Treatment5111.6 Follow-Up of Subjects with AEs5111.7 Pregnancy in the Clinical Study51 | 11. | 2 Monitoring for AEs | 48 |
| 11.5 Unmasking of the Study Treatment5111.6 Follow-Up of Subjects with AEs5111.7 Pregnancy in the Clinical Study51 | 11. | | |
| 11.5 Unmasking of the Study Treatment5111.6 Follow-Up of Subjects with AEs5111.7 Pregnancy in the Clinical Study51 | 11. | | |
| 11.6 Follow-Up of Subjects with AEs5111.7 Pregnancy in the Clinical Study51 | 11. | • | |
| 11.7 Pregnancy in the Clinical Study | | | |
| 12 ANALYSIS PLAN | | • | |

| Alcon - Bus<br>Document: TDO | mess ese only | <b>Date:</b> 08-Nov-2019 |
|---|---|---|
| Status: Effect | | Page <b>5</b> of <b>60</b> |
| 12.2 | Analysis Sets | 52 |
| 12.3 | Demographic and Baseline Characteristics | 52 |
| 12.4 | Effectiveness Analyses | 53 |
| | 12.4.1 Analysis of Primary Effectiveness Endpoint(s) | 53 |
| | 12.4.1.1 Statistical Hypotheses | 53 |
| | 12.4.1.2 Analysis Methods | |
| | 12.4.2 Analysis of Secondary Effectiveness Endpoints | |
| | 12.4.2.1 Statistical Hypotheses and Model | |
| 12.5 | 12.4.2.2 Analysis Methods | |
| 12.5 | Safety Analyses | |
| 12.7 | Interim Analyses and Reporting | |
| 12.7 | Sample Size Justification | |
| | ANDLING AND ADMINISTRATIVE REQUIREMENTS | |
| 13.1 | Subject Confidentiality | |
| 13.1 | Completion of Source Documents and Case Report Forms | |
| 13.2 | Data Review and Clarifications | |
| 13.4 | Sponsor and Monitoring Responsibilities | |
| 13.5 | Regulatory Documentation and Records Retention | |
| 13.6 | Quality Assurance and Quality Control | |
| | Quality Fissurance and Quality Condo | |
| | ENCES | |
| 15.1 | References Applicable for All Clinical Studies | 60 |
| | 15.1.1 US References Applicable for Clinical Studies | |
| 15.2 | Additional References for This Clinical Study | |
| | Link of Tables | |
| Table 2–1 | <b>List of Tables</b> List of Acronyms and Abbreviations Used in This Protocol | 11 |
| | · | |
| Table 3–1 | Schedule of Study Procedures and Assessments | 18 |
| Table 6–1 | Primary Objective(s) | 25 |
| Table 6–2 | Safety Objective(s) | 25 |

| Alcon - Busi | ness Use Only Pro | | | | Effective Date: 08-Nov-2019 | |
|---|---|---|---|---|---|---|
| Document: TDO | C-0056910 | Version: 2.0; | Most-Recent; Ef | fective; | | |
| Status: Effect: | ive | | | | Page <b>6</b> of <b>6</b> | 0 |
| Table 9–1 | Test Product | | | | 30 | 0 |
| Table 9–2 | Control Product. | | | | 33 | 3 |
| | | List of | Figures | | | |
| Figure 7-1 | Flowchart of Stu | dy Visits | | | 20 | 6 |
| Figure 11–1 | Categorization of | f All AEs | | | 4 | 5 |
| Figure 11–2 | Categorization or | f All SAE | | | 40 | 6 |


Status: Effective 

# 1 GLOSSARY OF TERMS

| Names of Test Product(s) | Throughout this document, test product(s) will be referred to as soft contact lenses or contact lenses |
|---|---|
| | Soft contact tenses of |
| Name of Control Product(s) | CooperVision® BIOFINITY® soft contact lenses (Biofinity |
| | contact lenses or Biofinity) |
| Adverse Device Effect | Adverse event related to the use of an investigational |
| (ADE) | medical device (test product) or control product. Note: This |
| | definition includes adverse events resulting from insufficient |
| | or inadequate instructions for use, deployment, |
| | implantation, installation, or operation; any malfunction; |
| | and use error or intentional misuse of the test product or |
| | control product. |
| Adverse Event (AE) | Any untoward medical occurrence, unintended disease or |
| | injury, or untoward clinical signs (including abnormal |
| | laboratory findings) in subjects, users or other persons, |
| | whether or not related to the investigational medical device |
| | (test product). <i>Note: For subjects, this definition includes</i> |
| | events related to the test product, the control product, or the |
| | procedures involved. For users or other persons, this |
| | definition is restricted to events related to the test product. |
| | Requirements for reporting Adverse Events in the study can |
| | be found in Section 11. |
| Anticipated Serious | Serious adverse device effect which by its nature, incidence, |
| Adverse Device Effect | severity, or outcome has been identified in the risk |
| | management file. |
| Device Deficiency | Inadequacy of a medical device with respect to its identity, |
| | quality, durability, reliability, safety, or performance. <i>Note:</i> |
| | This definition includes malfunctions, use errors, and |
| | inadequate labeling. |

Document: TDOC-0056910

Version: 2.0; Most-Recent; Effective; CURRENT

Status: Effective 

| | Degringments for more orting Desire Deficiencies in 11 11 |
|---|---|
| | Requirements for reporting Device Deficiencies in the study |
| | can be found in Section 11. |
| Enrolled Subject | Any subject who signs an informed consent form for |
| | participation in the study. |
| Interventional Clinical Trial | A research trial that prospectively assigns, whether |
| | randomly or not, human participants or groups of humans to |
| | one or more health-related interventions to evaluate the |
| | effects on health outcomes, and/or a research trial in which |
| | diagnostic or monitoring procedures beyond standard of care |
| | are conducted and generate outcomes for use in analysis of |
| | data. |
| Investigational Product | Is defined as a preventative (vaccine), a therapeutic (drug or |
| mvestigational i foduct | |
| | biologic), device, diagnostic, or palliative used as a test or |
| | control product in a clinical trial, including a product with a |
| | marketing authorization when used or assembled |
| | (formulated or packaged) in a way different from the |
| | authorized form, or when used for an unauthorized |
| | indication, or when used to gain further information about |
| | the authorized form. |
| Malfunction | Failure of a medical device to perform in accordance with its |
| | intended purpose when used in accordance with the |
| | instructions for use or clinical investigation plan. |
| Non-serious Adverse Event | Adverse event that does not meet the criteria for a serious |
| | adverse event. |
| Randomized Subjects | Any subject who is assigned a randomized treatment. |
| 3 | |
| Serious Adverse Device | Adverse device effect that has resulted in any of the |
| Effect (SADE) | consequences characteristic of a serious adverse event. |
| , | 1 |
| Serious Adverse Event | Adverse event that led to any of the following: |
| (SAE) | |
| | Death. |


Status: Effective 

• A serious deterioration in the health of the subject that either resulted in:

- a. a life-threatening illness or injury.

  Note: Life-threatening means that the individual was at immediate risk of death from the event as it occurred, ie, it does not include an event which hypothetically might have caused death had it occurred in a more severe form.
- b. any potentially sight-threatening event or permanent impairment to a body structure or a body function.
- c. in-patient hospitalization or prolonged hospitalization.

*Note: Planned hospitalization for a pre*existing condition, without serious deterioration in health, is not considered a serious adverse event. In general, hospitalization signifies that the individual remained at the hospital or emergency ward for observation and/or treatment (usually involving an overnight stay) that would not have been appropriate in the physician's office or an out-patient setting. Complications that occur during hospitalization are adverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious.

- d. a medical or surgical intervention to preventa) or b).
- e. any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use.


Status: Effective 

| | Fetal distress, fetal death, or a congenital abnormality or birth defect. Refer to Section 11 for additional SAEs. |
|---|---|
| Significant Non-Serious<br>Adverse Event | Is a symptomatic, device-related, non-sight threatening adverse event that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. |
| | Refer to Section 11 for additional Significant Non-Serious AEs. |
| Unanticipated Serious Adverse Device Effect | Serious adverse device effect which by its nature, incidence, severity, or outcome has not been identified in the risk management file. |
| Use Error | Act or omission of an act that results in a different medical device response than intended by manufacturer or expected by user. Note: This definition includes slips, lapses, and mistakes. An unexpected physiological response of the subject does not in itself constitute a use error. |


Status: Effective 

## 2 LIST OF ACRONYMS AND ABBREVIATIONS

Table 2-1 List of Acronyms and Abbreviations Used in This Protocol

| Abbreviation | Definition |
|---|---|
| ADE | Adverse device effect |
| AE | Adverse event |
| BCVA | Best corrected visual acuity |
| Biofinity contact | CooperVision BIOFINITY (comfilcon A) soft contact lenses |
| lens, Biofinity soft | |
| contact lens, or | |
| Biofinity | |
| CFR | Code of Federal Regulations |
| CLEAR CARE | CLEAR CARE Cleaning & Disinfecting Solution |
| COL | Clinical operations lead |
| CRF | Case report form |
| CSM | Clinical site manager |
| CTT | Clinical trial team |
| D | Diopter(s) |
| D/C | Discontinue |
| eCRF | Electronic case report form |
| EDC | Electronic data capture |
| FDA | US Food and Drug Administration |
| GCP | Good Clinical Practice |
| IB | Investigator's brochure |
| ICF | Informed consent form |
| ICH | International Council for Harmonisation of Technical |
| | Requirements for Pharmaceuticals for Human Use |
| IEC | Independent ethics committee |
| IP | Investigational product |
| IRB | Institutional review board |
| IRT | Interactive response technology |
| ISO | International Organization for Standardization |
| LID | Lens identification |
| logMAR | Logarithm of the minimum angle of resolution |
| mm | Millimeter |
| MOP | Manual of procedures |
| N/A | Not applicable |
| contact lens | soft contact lenses |
| or | |
| OD | Right eye |
| OS | Left eye |
| OU | Both eyes |


Status: Effective 

| Abbreviation | Definition |
|--------------|-------------------------------|
| SAE | Serious adverse event |
| SADE | Serious adverse device effect |
| SiHy | Silicone hydrogel |
| SOP | Standard operating procedure |
| US/USA | United States of America |
| USAN | United States Adopted Name |
| USV | Unscheduled visit |
| VA | Visual acuity |
| VS | Versus |


Status: Effective 

## 3 PROTOCOL SUMMARY

| This will be a prospective, randomized, | | controlled |
|-----------------------------------------|--------------------|------------|
| double-masked, parallel-group daily we | ar clinical study. | - |

Approximately 8 sites in the US will enroll approximately 120 subjects. Subjects will be expected to attend 6 office visits: Screening/Baseline/Dispense, Week 1 Follow-up, Week 2 Follow-up, Month 1 Follow-up, Month 2 Follow-up, and Month 3 Follow-up/Exit. The total expected duration of participation for each subject is approximately 3 months in this daily wear clinical study. Approximately 80 subjects will be assigned to wear the test lenses and 40 subjects will be assigned to wear the control lenses, following the 2:1 subject allocation ratio as recommended by ISO 11980:2012 and the US FDA 510(k) guidance document.

| Subjects and the study personnel conducting the study evaluations will be masked to |
|---|
| treatment. Subjects who meet the inclusion and exclusion criteria will be randomized to wear |
| either the test contact lenses in both eyes or the control contact lenses (Biofinity) in |
| both eyes for 3 months of daily wear exposure. Following randomization, subjects will be |
| trial fit in the assigned study lens using the fitting set supplied by the Sponsor, and the overall |
| fit and correct contact lens power for each eye will be determined. |
| The delegated staff |
| member will then complete a contact lens order form to obtain lenses for each subject. The |
| Sponsor will send investigational products for each subject to the site after receiving an order |
| from the Investigator. |

At the Screening/Baseline/Dispense Visit, study lenses will be dispensed to qualified subjects and the subject will be provided with sufficient lens supplies to follow a monthly replacement schedule until the next visit. All study lenses will be worn for at least 5 days per week and 8 hours per day in a daily wear modality (eg, will not be worn while sleeping).

Problem lenses (if any) will not be discarded, but collected by the subject and returned to the investigational site. Regardless of whether the subject is randomized to the test or the control group, CLEAR CARE® Cleaning & Disinfecting Solution (CLEAR CARE) must be used for cleaning and disinfection.


Status: Effective 

Visual acuity with study lenses will be measured at all visits, and any decrease of 2 or more lines from the Screening/Baseline/Dispense Visit to any follow-up visit should be explained by the Investigator.

| Investigational | Medical Device |
|---|---|
| Product Type | |
| Study Type | Interventional |
| Investigational | Test Product: soft contact lens |
| Products | Control Product: Biofinity soft contact lens |
| Purpose and | The purpose of this clinical study is to evaluate the performance of |
| Rationale | the investigational soft contact lens compared to the |
| | commercially available Biofinity soft contact lens when worn in a |
| | daily wear modality, by assessing visual acuity as the primary |
| | variable. |
| | The overall objective is to evaluate safety and effectiveness of the |
| | soft contact lens when worn for daily wear and replaced |
| | monthly as compared to Biofinity soft contact lens. |
| | monthly as compared to Biolimity soft contact lens. |
| Objective(s) | The primary objective is to evaluate visual acuity of the |
| | investigational soft contact lens compared to the |
| | commercially available Biofinity soft contact lens. |
| Endpoint(s) | Primary Effectiveness |
| | Distance VA (Snellen) with study lenses |


Status: Effective 

| • | AEs |
|-----------------|--------------------------------------------------|
| | Biomicroscopy findings |
| | D : 1 C : : |
| Assessment(s) I | Effectiveness |
| | VA with study lenses (Snellen distance) |
| • | VA with habitual correction (Snellen distance) |
| • | Manifest refraction |
| | BCVA (Snellen distance with manifest refraction) |


Status: Effective 

| | <ul> <li>Discontinuations with reason</li> <li>Safety</li> <li>AEs</li> <li>Biomicroscopy</li> <li>Device deficiencies</li> </ul> |
|---|---|
| Study Design | This will be a prospective, randomized, controlled, double-masked, parallel-group, daily wear clinical study. Subject participation in the study will be approximately 14 weeks with approximately 3 months of exposure to study lenses. |
| Subject Population | Volunteer subjects aged 18 or over who are adapted daily wear frequent replacement soft contact lens wearers, excluding Biofinity habitual wearers, have at least 3 months of soft contact lens wearing experience, and who wear their habitual lenses at least 5 days per week and at least 8 hours per day. Subjects must require contact lens correction in a sphere power range from -1.00 to -6.00 D. |


Status: Effective 

| Key Inclusion Criteria (See Section 8.1 for a complete list of inclusion criteria) Key Exclusion Criteria (See Section 8.2 for a complete list of exclusion criteria) Data Analysis and Sample Size Justification | <ul> <li>Successful wear of spherical daily wear frequent replacement soft contact lenses for distance correction in both eyes during the past 3 months for a minimum of 5 days per week and 8 hours per day.</li> <li>Manifest cylinder ≤ 0.75 D in each eye</li> <li>Wearing habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment.</li> <li>Monovision contact lens wearers</li> <li>Habitually wearing Biofinity lenses</li> <li>In adherence to the reporting format as specified in the ISO clinical standard and FDA 510(k) guidance documents, effectiveness and safety data will be presented separately based upon subject study status of Completed or Discontinued.</li> <li>No formal hypotheses are formulated for the primary effectiveness endpoint; hence, no inferential testing will be performed.</li> <li>Descriptive statistics will be provided on the Snellen categories as well as the converted logMAR values. Similarly, all supportive endpoints will be summarized descriptively according to each measurement scale.</li> <li>Sample size is based upon ISO clinical standard and FDA 510(k) requirements with the recommendations of at least 50 subjects in the Test group, in a 2:1 Test to Control ratio.</li> </ul> |
|---|---|
| Key Words | Biofinity, daily wear, registration |
| Associated Materials | CLEAR CARE will be used for daily cleaning and disinfection. |

Table 3-1 Schedule of Study Procedures and Assessments

| Procedure/ Assessment | Visit 1<br>Screening/<br>Baseline/<br>Dispense | Visit 2<br>Week 1<br>Follow-up <sup>5</sup> | Visit 3<br>Week 2<br>Follow-up <sup>5</sup> | Visit 4<br>Month 1<br>Follow-up <sup>5</sup> | Visit 5<br>Month 2<br>Follow-up <sup>5</sup> | Visit 6<br>Month 3<br>Follow-<br>up/Exit <sup>5</sup> | Early<br>Exit | USV |
|---|---|---|---|---|---|---|---|---|
| | Day 1 | Day 8<br>(-2/+2 days) | Day 15<br>(-3/+3 days) | Day 30<br>(-3/+5<br>days) | Day 60<br>(-3/+5<br>days) | Day 95<br>(-3/+5<br>days) | | |
| Informed Consent | X | | | | | | | |
| Demographics | X | | | | | | | |
| Medical History | X | X | X | X | X | X | X | (X) |
| Concomitant Medications | X | X | X | X | X | X | X | (X) |
| Inclusion/Exclusion | X | | | | | | | |
| Habitual lens information<br>(brand/manufacturer, power, modality/wear<br>success, habitual lens care brand) | X | | | | | | | |
| VA w/ habitual correction (OD,OS<br>Snellen distance) | X | | | | | X | X | (X) |
| Manifest refraction <sup>4</sup> | X | (X) | (X) | (X) | (X) | X | X | (X) |
| BCVA <sup>4</sup> (OD,OS Snellen distance with manifest refraction) | X | (X) | (X) | (X) | (X) | X | X | (X) |
| Biomicroscopy | X | X | X | X | X | X | X | (X) |

Alcon - Business Use Only Protocol - Clinical Document: TDOC-0056910 Version: 2.0; Mo Status: Effective

| Procedure/ Assessment | Visit 1<br>Screening/<br>Baseline/<br>Dispense | Visit 2<br>Week 1<br>Follow-up <sup>5</sup> | Visit 3<br>Week 2<br>Follow-up <sup>5</sup> | Visit 4 Month 1 Follow-up <sup>5</sup> | Visit 5<br>Month 2<br>Follow-up <sup>5</sup> | Visit 6<br>Month 3<br>Follow-<br>up/Exit <sup>5</sup> | Early<br>Exit | USV |
|---|---|---|---|---|---|---|---|---|
| | Day 1 | Day 8<br>(-2/+2 days) | Day 15<br>(-3/+3 days) | Day 30<br>(-3/+5<br>days) | Day 60<br>(-3/+5<br>days) | Day 95<br>(-3/+5<br>days) | | |
| | X | | | | | | | |
| Randomize and record lens power | X | | | | | | | |
| | X | | | | | | | |
| Order study lenses* | X | | | | | | | |
| IP Dispense* | X | X | (X) | (X) | (X) | | | (X) |
| VA w/ study lenses<br>(OD, OS Snellen distance) <sup>1</sup> | X | X | X | X | X | X | X | (X) |

Print Date:

Alcon - Business Use Only Protocol - Clinical Document: TDOC-0056910 Version: 2.0; Mo Status: Effective

| Procedure/ Assessment | Visit 1<br>Screening/<br>Baseline/<br>Dispense | Visit 2<br>Week 1<br>Follow-up <sup>5</sup> | Visit 3<br>Week 2<br>Follow-up <sup>5</sup> | Visit 4 Month 1 Follow-up <sup>5</sup> Day 30 | Visit 5 Month 2 Follow-up <sup>5</sup> Day 60 | Visit 6 Month 3 Follow- up/Exit <sup>5</sup> Day 95 | Early<br>Exit | USV |
|---|---|---|---|---|---|---|---|---|
| | Day 1 | Day 8<br>(-2/+2 days) | Day 15<br>(-3/+3 days) | (-3/+5<br>days) | (-3/+5<br>days) | (-3/+5<br>days) | | |
| AE | v | v | v | v | v | v | v | (V) |
| AEs | X | X | X | X | X | X | X | (X) |
| Device deficiencies | X | X | X | X | X | X | X | (X) |
| Exit Form | (X) | (X) | (X) | (X) | (X) | X | X | (X) |

Print Date:

USV = Unscheduled Visit

\*source only <sup>5</sup>All follow-up visits should be scheduled at least 4 hours after lens insertion.

ct.


Status: Effective 

#### 4 PROTOCOL AMENDMENTS

Modification of the protocol is prohibited without prior written agreement in the form of a protocol amendment. All amendments must be created by the Study Sponsor and must be approved by the IRB/IEC and global and regional Health Authorities, as applicable, prior to implementation except when required to mitigate immediate safety risks or when the changes involve only logistical or administrative revisions.

Amendments may necessitate that the informed consent and other study-related material be revised. If the consent form is revised, all subjects currently enrolled in the study must sign the approved, revised informed consent (re-consent), as required by the IRB/IEC.

#### 4.1 Amendments

Amendment 1




Status: Effective 

#### 5 INTRODUCTION

## 5.1 Rationale and Background

Daily wear contact lenses are worn during waking hours for a full day, and then removed for cleaning and disinfection prior to reinsertion the following day. Frequent replacement daily wear contact lenses are replaced according to the product package insert provided by the contact lens manufacturer.



# 5.2 Purpose of the Study

The purpose of this clinical study is to evaluate the safety and performance of the investigational soft contact lens compared to the commercially available Biofinity soft contact lens when worn in a daily wear modality, by assessing VA as the primary variable.

At the end of the study, a clinical study report will be prepared in accordance with applicable regulatory requirements and standards.

Effective Date: 08-Nov-2019 Alcon - Business Use Only Protocol - Clinical Version: 2.0; Most-Recent; Effective; CURRENT **Document:** TDOC-0056910  Status: Effective There are no immediate plans to submit the results of this study for publication **Risks and Benefits** Contact lenses may offer improved peripheral vision and the convenience of not wearing spectacles. Material properties and design characteristics of contact lenses are features consistent with successful contact lens wear. Based upon nonclinical testing and documented rationale for applicability of test results, contact lenses are assessed to be non-toxic and biocompatible for on-eye use. In the US, Biofinity contact lenses have approved indications for use for both daily wear and extended wear for up to 6 continuous nights. Further details on any known potential risks and benefits can be found in the product package insert. A summary of the known potential risks and benefits associated with contact lenses can be found in the IB. The potential harms associated with on-eye exposure to the new lens materials include toxicity response, blurred vision, and ocular discomfort. In general, when worn for daily wear, the risks with contact lenses are anticipated to be similar to other marketed soft contact lenses worn for daily wear. There may also be unknown risks to the use of contact lenses. Any risk to subjects in this clinical study will be minimized by compliance with the eligibility criteria and study

There may also be unknown risks to the use of contact lenses. Any risk to subjects in this clinical study will be minimized by compliance with the eligibility criteria and study procedures, clinical oversight, and monitoring. Site personnel will educate subjects on proper hygiene, lens handling, and compliance with the use of contact lenses for daily wear according to the protocol. Subjects should be instructed not to wear contact lenses while swimming due to increased risk of infection or while sleeping. Site personnel should advise the subjects to remove contact lenses and return for prompt follow-up of symptoms such as ocular discomfort, foreign body sensation, excessive tearing, vision changes, or hyperemia.

Refer to the IB for additional information.


Status: Effective 

## **6 STUDY OBJECTIVES**

# 6.1 Primary Objective(s)

Table 6–1 Primary Objective(s)

| Objective(s) | Endpoint(s) |
|---|---|
| Evaluate VA of the investigational | Primary Effectiveness |
| soft contact lens compared to the commercially available Biofinity soft contact lens. | • Distance VA (Snellen) with study lenses |

## **6.2** Secondary Objective(s)

Not Applicable.

# 6.3 Exploratory Objective(s)

Not Applicable.

# 6.4 Safety Objective(s)

Table 6–2 Safety Objective(s)

| Objective(s) | Endpoint(s) |
|-----------------------------------------------|------------------------|
| Duty of care and evaluation of safety profile | AEs |
| of the investigational products. | Biomicroscopy findings |
| | Device deficiencies |

## 7 INVESTIGATIONAL PLAN

# 7.1 Study Design

This will be a prospective, randomized, controlled, double-masked, parallel-group, daily wear clinical study.

This clinical study will engage approximately 8 clinic sites to enroll approximately 120 subjects with approximately 15 subjects per site.


Status: Effective 

Subjects will be expected to attend 6 office visits: Screening/Baseline/Dispense, Week 1 Follow-up, Week 2 Follow-up, Month 1 Follow-up, Month 2 Follow-up, and Month 3 Follow-up/Exit. The total expected duration of participation for each subject is approximately 14 weeks with approximately 3 months of exposure to study lenses in this daily wear study. Subjects will be randomized to wear either the test contact lenses in both eyes or the control Biofinity contact lenses in both eyes.

Following randomization, study lenses will be dispensed to the subject. Subjects will be provided with sufficient lens supplies to follow a monthly replacement schedule until the next scheduled visit.

Subjects will wear the lenses while awake in a daily wear modality. CLEAR CARE will be used for daily cleaning and disinfection.

The estimated time to recruit subjects for this study is approximately 6 weeks. The study is expected to take approximately 14 weeks for completion from the last patient first visit. The study outline is provided below:

Figure 7-1 Flowchart of Study Visits




Status: Effective 

## 7.2 Rationale for Study Design

In this clinical study, the safety and performance of the investigational contact lens will be compared to the commercially available Biofinity contact lens in a double-masked, parallel-group design with approximately 3 months of daily wear exposure. The study is designed following the recommendations for registration from ISO 11980:2012 and the US FDA 510(k) daily wear contact lens guidance document.

## 7.3 Rationale for Duration of Treatment/Follow-Up

The duration of exposure and follow-up duration are in compliance with the recommended guidance from ISO 11980:2012.

#### 7.4 Rationale for Choice of Control Product

The Biofinity contact lens was chosen as the control product because this lens is a proper predicate device to compare to contact lens with regard to effectiveness and safety. Both the contact lens and Biofinity contact lens are monthly replacement SiHy lenses and are to be prescribed for daily wear. The Biofinity contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes. The lenses are intended to be cleaned and disinfected daily when worn for daily wear.

# 7.5 Data Monitoring Committee

Not Applicable.

#### 8 STUDY POPULATION

The study population consists of adult male or female subjects (aged 18 or over), with non-diseased eyes, who require optical correction for refractive ametropia (myopia and hyperopia). The aim is to enroll approximately 120 subjects at approximately 8 US sites, with approximately 15 subjects per site. Estimated time needed to recruit subjects for the study is approximately 6 weeks.

The intended study population consists of volunteer subjects who are frequent replacement daily wear soft contact lens wearers, excluding Biofinity habitual wearers, who have at least 3 months of contact lens wearing experience, and who wear their habitual lenses at least 5 days per week and 8 hours per day.


Status: Effective 

#### 8.1 Inclusion Criteria

Written informed consent must be obtained before any study specific assessment is performed. Upon signing informed consent, the subject is considered enrolled in the study.

Subjects eligible for inclusion in this study must fulfill all of the following criteria:

- 1. At least 18 years of age.
- 2. Able to understand and sign an IRB/IEC approved Informed Consent form.
- 3. Willing and able to attend all scheduled study visits as required per protocol.
- Successful wear of spherical daily wear frequent replacement soft contact lenses for distance correction in both eyes during the past 3 months for a minimum of 5 days per week and 8 hours per day.
- 5. Manifest cylinder  $\leq 0.75$  D in each eye.
- 6. Best spectacle corrected (using manifest refraction) VA 20/25 or better in each eye.
- 7. Requiring contact lens sphere power from -1.00 to -6.00 D and willing to wear assigned study lenses as required per protocol
- Distortion-free keratometric readings.



 Possess and willing to wear habitual spectacles for vision correction when study lenses are not worn, if needed.


Status: Effective 

#### 8.2 Exclusion Criteria

Subjects fulfilling any of the following criteria are not eligible for participation in this study.

1. Any anterior segment infection, inflammation, or abnormality or disease (including systemic) that contraindicates contact lens wear, as determined by the Investigator.

- 2. Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the Investigator.
- 3. History of ocular or intraocular surgery, including refractive surgery, and/or irregular cornea;
- 4. Current or previous orthokeratology treatment or has worn rigid gas permeable lenses in the past 12 months.
- 5. Biomicroscopy findings at screening that are moderate (Grade 3) or higher and/or corneal vascularization that is mild (Grade 2) or higher; presence of corneal infiltrates.
- 6. Current or history of pathologically dry eye in either eye that, in the opinion of the Investigator, would preclude contact lens wear.
- 7. Current or history of herpetic keratitis in either eye.
- 8. Eye injury in either eye within 12 weeks immediately prior to enrollment for this study.
- 9. Current or history of intolerance, hypersensitivity, or allergy to any component of study lenses, lens care or associated materials for the study.
- 10. Wearing daily disposable lenses over the last 3 months prior to enrollment.
- 11. No prior experience with routine cleaning and disinfection.
- 12. Wearing habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment.
- 13. Any use of habitual/prescribed topical ocular medications or artificial tear or rewetting drops (habitual) that would require instillation during study lens wear.
- 14. Monovision or multifocal contact lens wearers.


Status: Effective 

15. The Investigator, his/her staff, family members of the Investigator, family members of the Investigator's staff, or individuals living in the households of the aforementioned persons may not participate in the study.

- 16. Participation of the subject in a clinical study within the previous 30 days or currently enrolled in any clinical study.
- 17. Any habitual wear of Biofinity contact lenses.

Women of childbearing potential or women who are pregnant at the time of study entry are not excluded from participation. Pregnancy should be included in the Medical History section of the eCRF when a pregnant woman enters the study or if a woman becomes pregnant during the study. Pregnancy is not reportable as an AE; however, complications may be reportable and will be decided on a case-by-case basis.

## 8.3 Rescreening of Subjects

Rescreening of subjects is not allowed in this study.

#### 9 TREATMENTS ADMINISTERED

## 9.1 Investigational Product(s)

Test Product(s): soft contact lenses

Control Product(s) (If applicable): Biofinity (comfilcon A) soft contact lenses

Table 9–1 Test Product

| Test Product | soft contact lenses contact lens) |
|--------------|-----------------------------------|
| | (LID018869) |
| Manufacturer | Alcon |
| | 6201 South Freeway |
| | Fort Worth, Texas 76134-2099 |
| | USA |


Status: Effective 

| Status: Effective | 1 age 31 01 00 |
|---|---|
| Indication for Use and Intended Purpose in the Current Study | The intended use of this contact lens is for vision correction. |
| Product Description<br>and Parameters<br>Available for this<br>Study | <ul> <li>Water content target: 55 ± 2%</li> <li>Power range: -1.00 to -6.00 D (0.25 D steps)</li> <li>Base curve: 8.4 mm (±0.2 mm)</li> <li>Diameter: 14.2 mm (±0.2 mm)</li> </ul> |
| Formulation | Silicone hydrogel. Additional details can be found in the IB. |
| Usage | <ul> <li>Wear: <ul> <li>During waking hours only.</li> <li>Subjects will wear a fresh pair of lenses in alignment with monthly planned replacement schedule.</li> <li>Bilateral</li> </ul> </li> <li>Exposure: At least ~8 hours per day and ~5 days per week over ~3 month's exposure period.</li> <li>Replacement period: Monthly planned replacement over the course of the study duration. <ul> <li>Monthly replacement for this trial is defined as 27 – 35 days.</li> <li>For planned replacement, lenses will be replaced even if one or both of the lenses have not been used for the full month wearing schedule.</li> </ul> </li> <li>Lens Care: CLEAR CARE (mandatory).</li> <li>Additional details can be found in the MOP.</li> </ul> |


Status: Effective 

| Number/Amount of | At each study visit, sites will ensure that subjects are given adequate |
|---|---|
| Product to be | lenses to last until the next planned study visit, allowing for planned |
| Provided to the | and unplanned lens replacements. |
| Subject | |
| Packaging | Blister foil pack |
| Description | |
| Labeling | Lens Foil label includes: |
| Description | - identifier |
| | - base curve |
| | - diameter |
| | - manufacturing protocol number |
| | - packing solution |
| | - power |
| | - lot number |
| | - expiration date |
| | - content statement |
| | - investigational device statement |
| | - Sponsor information |
| | • Provided in packages of approximately 6, identified with the following: |
| | - a color-coded label stating the protocol number |
| | - identifier |
| | - power |
| | - an investigational use only statement |
| | - tracking number |
| Storage Conditions | Stored at room temperature. |


Status: Effective 

| Supply | • Fitting sets will be provided by the Sponsor before the start of the study to be used during Visit 1. The site will dispense the study lenses to the subject at Visit 1 from the fitting set. Fitting sets will be resupplied, as needed. |
|---|---|
| | • Based on the Investigator's lens order form, the Sponsor will send study lenses (as well as spare lenses) to the site for each subject. The site will provide the study lenses to the subject at Visit 2, and at subsequent follow-up visits, as needed, to allow for both planned lens replacement schedule and any unplanned lens replacements throughout the study. Refer to the MOP for a detailed description. |

## Table 9–2 Control Product

| Control Product(s) | Biofinity (comfilcon A) soft contact lenses (Biofinity contact lens) (LID010221) |
|---|---|
| Manufacturer | CooperVision |
| Indication for Use | The intended use of this contact lens is for vision correction. |
| Product Description<br>and Parameters<br>Available for this<br>Study | <ul> <li>Material: comfilcon A</li> <li>Water content: 48%</li> <li>Power range: -1.00 to -6.00 D (0.25 D steps)</li> <li>Base curve: 8.6 mm</li> <li>Diameter: 14.0 mm</li> </ul> |
| Formulation | Silicone Hydrogel. Additional details can be found in the Biofinity package insert. |
| Usage | <ul> <li>Wear:</li> <li>Daily Wear</li> <li>During waking hours only.</li> </ul> |


| Status: Effective | | | | | | | Page <b>34</b> of <b>60</b> |
|---|---|---|---|---|---|---|---|
| | O 1 ' | .11 | C | 1 | • | C 1 | • |

| | <ul> <li>Subjects will wear a fresh pair of lenses in<br/>alignment with monthly planned replacement<br/>schedule.</li> </ul> |
|---|---|
| | o Bilateral |
| | • Exposure: At least ~8 hours per day and ~5 days per week over ~3 month's exposure period. |
| | Replacement period: Monthly planned replacement over the course of the study duration. |
| | <ul> <li>Monthly replacement for this trial is defined as 27 –</li> <li>35 days.</li> </ul> |
| | <ul> <li>For planned replacement, lenses will be replaced even if<br/>one or both of the lenses have not been used for the full<br/>month wearing schedule.</li> </ul> |
| | Lens Care: CLEAR CARE (mandatory), |
| | Additional details can be found in the MOP. |
| Number/Amount of | At each study visit, sites will ensure that subjects are given adequate |
| Product to be | lenses to last until the next planned study visit, allowing for planned |
| Provided to the Subject | and unplanned lens replacements. |
| Packaging Description | Blister foil pack. |
| Labeling | Lens Foil label includes: |
| Description | - identifier |
| | - base curve |
| | - diameter |
| | - packing solution |
| | - power |
| | - lot number |
| | - expiration date |


Status: Effective 

| | - content statement |
|---|---|
| | - investigational device statement |
| | - Sponsor information |
| | • Provided in packages of approximately 6, identified with the following: |
| | - a color-coded label stating the protocol number |
| | - identifier |
| | - power |
| | - an investigational use only statement |
| | - tracking number |
| Storage Conditions | Stored at room temperature. |
| Supply | • Fitting sets will be provided by the Sponsor before the start of the study to be used during Visit 1. The site will dispense the study lenses to the subject at Visit 1 from the fitting set. Fitting sets will be resupplied, as needed. |
| | • Based on the Investigator's lens order form, the Sponsor will send study lenses (as well as spare lenses) to the site for each subject. The site will provide the study lenses to the subject at Visit 2, and at subsequent follow-up visits, as needed, to allow for both planned lens replacement schedule and any unplanned lens replacements throughout the study. Refer to the MOP for a detailed description. |

More information on the test product can be found in the IB; information on the control product can be found in the Package Insert.

# 9.2 Other Medical Device or Medication Specified for Use During the Study

Other than the pre-specified CLEAR CARE, LacriPure (or equivalent), and Systane rewetting drops, no other ocular medical devices or medications are allowed to be used during the clinical study.


Status: Effective 

## 9.3 Treatment Assignment/Randomization



Only after signing the ICF, a subject will be assigned a subject number by the electronic data capture system.

A randomization list will be generated using a validated system that automates the random assignment of treatment arms to randomization numbers in the specified ratio

Subjects will be assigned a treatment arm according to the randomization list uploaded in the IRT system. The randomization list will be generated and maintained by the Study Sponsor.

At Visit 1, all eligible subjects will be randomized via the EDC/IRT integration system to one of the treatment arms. The Investigator's delegate will access the respective system after confirming that the subject meets all the eligibility criteria. A randomization number will be automatically assigned to the subject according to the subject randomization list but will not be communicated to the site user. The EDC/IRT integration system will inform the site user of the treatment assignment to be dispensed to the subject.

# 9.4 Treatment Masking

This study is double-masked, with subjects randomized to use or Biofinity contact lenses for the duration of the 3-month treatment period. All members associated with the study (at the site and the Study Sponsor) will be masked to the assigned treatment



Status: Effective 

| Status. Effective | 1 age 37 of 00 |
|-------------------|----------------|


Status: Effective 



This level of masking will be maintained throughout the conduct of the study. Unmasking will occur only after all planned study data have been validated, and the database locked.

Masked study personnel must avoid seeking information that may compromise masking.



In the event of a medical emergency where the knowledge of subject treatment is required, individual Investigator(s) will have the ability to unmask the treatment assignment for a specific subject. If time allows, the appropriate Study Sponsor representative should be contacted prior to unmasking. Unmasking must be done according to the instructions provided for the study IRT system.

# 9.5 Accountability Procedures

Upon receipt of the IPs, the Investigator or delegate must conduct an inventory. During the study, designated study staff must provide the IPs to the subjects in accordance with their randomization assignment. Throughout the study, the designated study staff must maintain records of IP dispensation and collection for each subject. This record must be made available to the study monitor for the purposes of verifying the accounting of IP supplies. Any discrepancies and/or deficiencies between the observed disposition and the written account must be recorded along with an explanation. All IPs sent to the Investigator must be accounted for by Study Sponsor personnel, and in no case be used in an unauthorized situation.


Status: Effective 

It is the Investigator's responsibility to ensure that:

All study products are accounted for and not used in any unauthorized manner

- All used foils and unused supplies are returned by each subject
- All unused products are available for return to the Study Sponsor, as directed
- Any study lenses associated with a device deficiency or with any product-related AE (ie, ADE or SADE) are returned to the Study Sponsor for investigation, unless otherwise directed by the Sponsor. Refer to Section 11 of this protocol for additional information on the reporting of device deficiencies and AEs and the MOP for the return of study products associated with these events.

The Investigator is responsible for proper disposition of all unused IPs at the conclusion of the study, according to the instructions provided in the MOP.

## 9.6 Changes to Concomitant Medications, Treatments/Procedures

After the subject is enrolled into the study, the Investigator must instruct the subject to notify the study site about:

- Any new medications
- Alterations in dose or dose schedules for current medications
- Any medical procedure or hospitalization that occurred or is planned
- Any non-drug therapies (including physical therapy and blood transfusions)

The Investigator must document this information in the subject's case history source documents

#### 10 STUDY PROCEDURES AND ASSESSMENTS

Subjects will be expected to attend 6 office visits, as shown below.

| Visit # | Visit Type | Visit Day | Visit Window |
|---|---|---|---|
| Visit 1 | Screening/Baseline/Dispense | Day 1 | N/A |
| Visit 2 | Week 1 Follow-up Visit | Day 8 | Days 6-10 |
| Visit 3 Week 2 Follow-up Visit | | Day 15 | Days 12–18 |
| Visit 4 | Month 1 Follow-up Visit | Day 30 | Days 27–35 |


Status: Effective 

| Visit # | Visit Type | Visit Day | Visit Window |
|---------|------------------------------|-----------|--------------|
| Visit 5 | Month 2 Follow-up Visit | Day 60 | Days 57–65 |
| Visit 6 | Month 3 Follow-up/Exit Visit | Day 95 | Days 92–100 |

Unscheduled Visits and Early Termination Visits are allowed, if necessary.

At the Screening/Baseline/Dispense Visit, following randomization, assigned study lenses will be trial fit using the fitting sets supplied by the Sponsor, and the overall fit and correct contact lens power for the individual subject will be determined. Sites will be provided with an adequate lens supply to dispense the first pair of study lenses during Visit 1 to qualified subjects according to the randomization schedule.

| At the Screening/Baseline/Dispense Visit, study lenses will be dispensed to the subject. All subjects will wear the study lenses in a daily wear modality, only during waking hours. |
|---|
| Subjects assigned to wearing or Biofinity contact lenses will insert a new pair of lenses each month and discard them at the end of the month. Problem lenses (if any) will no |
| be discarded, but collected by the subject and returned to the investigational site. |
| . VA with study lenses will be measured at all visits, and any decrease of 2 or |
| more lines from the Screening/Baseline/Dispense Visit to any follow-up visit should be |
| explained by the Investigator. |

# 10.1 Informed Consent and Screening

The Investigator or delegate must explain the purpose and nature of the study, and have the subject read, sign, and date the IRB/IEC-approved informed consent document. The subject must sign the ICF BEFORE any study-specific procedures or assessments can be performed, including study-specific screening procedures. Additionally, have the individual obtaining consent from the subject and a witness, if applicable, sign and date the informed consent document.


Status: Effective 

The Investigator or delegate must provide a copy of the signed document to the subject and place the original signed document in the subject's chart, or provide documentation as required by local regulations.

## **10.2 Description of Study Procedures and Assessments**

Detailed descriptions of assessments and procedures are provided in the MOP. The Investigator is responsible for ensuring responsibilities for all procedures and assessments are delegated to appropriately qualified site personnel.

## 10.2.1 Demographics

Obtain demographic information including age, race, ethnicity, and sex.

## 10.2.2 Medical History

Collect medical history information, including information on all medications used within the past 30 days. Include herbal therapies, vitamins, and all over-the-counter as well as prescription medications. Throughout the subject's participation, obtain information on any changes in medical health and/or the use of concomitant medications.

## 10.2.3 Investigational Product Compliance

Review subject compliance with the IP usage and adjunct product usage and collect all used and unused study IPs and other products that were dispensed.

# 10.2.4 Adverse Event Collection: Safety Assessment

Assess and record any AEs that are observed or reported, including those associated with changes in concomitant medication dosing since the previous visit. Requirements for reporting AEs in the study can be found in Section 11.

# 10.2.5 Slit-Lamp Biomicroscopy: Safety Assessment

A slit-lamp examination must be performed in both eyes before instillation of any diagnostic eye drops.

# 10.2.6 Device Deficiencies: Safety Assessment

Assess and record any device deficiencies that are reported or observed, since the previous visit. Requirements for reporting device deficiencies in the study can be found in Section 11.


Status: Effective 

## 10.2.7 Visual Acuity: Effectiveness Assessment



Refer to the MOP for additional details.

## **10.3 Additional Study Assessments**

Additional effectiveness assessments will be conducted throughout the course of the study for. Refer to the MOP for details on each of these assessments.

Refer to Table 3–1.

#### 10.4 Unscheduled Visits

If a subject visit occurs between any regularly scheduled visits, this visit must be documented as an Unscheduled Visit or Early Exit as applicable. During all unscheduled visits, the Investigator must conduct the following procedures, as appropriate:

- Collect AE information, as applicable
- Record changes in medical condition or concomitant medication, as applicable
- Collect device deficiency information, as applicable
- VA with habitual correction
- Manifest refraction
- BCVA with manifest refraction

- Perform biomicroscopy (assessments with or without lenses, as applicable)
- VA with study lenses

Alcon - Business Use Only Protocol - Clinical Effective Date: 08-Nov-2019


Status: Effective 

The Investigator may perform additional procedures for proper diagnosis and treatment of the subject according to Table 3–1. The Investigator must document this information in the subject's case history source documents.

If, during an Unscheduled Visit, the subject is to discontinue IP or is discontinuing from the study, the Investigator must conduct Exit procedures according to Table 3–1, as possible. Do not complete an Unscheduled Visit if a subject is exiting between scheduled study visits. An Early Exit assessment should be completed instead.

## 10.5 Discontinued Subjects

#### 10.5.1 Screen Failures

Screen failures are subjects who were excluded from the study after signing the informed consent, not meeting the inclusion/exclusion criteria, and prior to randomization to product/dispense of study product.

The Investigator must document the reason for screen failure in the subject's case history source documents.

Subject numbers must not be re-used.

#### 10.5.2 Discontinuations

Discontinued subjects are individuals who voluntarily withdraw or are withdrawn from the study by the Investigator after signing the informed consent.

Subject numbers of discontinued subjects must not be re-used.

Subjects may discontinue from study or study treatment at any time for any reason. Subjects may also be discontinued from study treatment at any time if, in the opinion of the Investigator, continued treatment poses a risk to their health.


Status: Effective 

For subjects discontinuing from the study, the Investigator must complete all Exit procedures according to Table 3–1, if the subject is willing and able, and if in the opinion of the Investigator it is safe for the subject to do so.

The Investigator must document the reason for study or treatment discontinuation in the subject's case history source documents.

To ensure the safety of all subjects who discontinue early, Investigators must assess each subject and, if necessary, advise them of any therapies and/or medical procedures that may be needed to maintain their health.

# 10.5.3 Schedule of Procedures and Assessments for Subjects Discontinued from Investigational Product

Other than screen failures, if a subject discontinues from the study, the subject should undergo an Early Exit Visit. Refer to Table 3–1.

#### 10.6 Clinical Study Termination

The Study Sponsor reserves the right to close the investigational site or terminate the study in its entirety at any time.

If the clinical study is prematurely terminated or suspended by the Study Sponsor:

- The Study Sponsor must:
  - Immediately notify the Investigator(s) and subsequently provide instructions for study termination.
  - Inform the Investigator and the regulatory authorities of the termination/suspension and the reason(s) for the termination/suspension.
- The Investigator must:
  - Promptly notify the IRB/IEC of the termination or suspension and of the reasons.
  - Provide subjects with recommendations for post-study treatment options as needed.

The Investigator may terminate the site's participation in the study for reasonable cause.


Status: Effective 

## 10.6.1 Follow-up of Subjects After Study Participation Has Ended

Following this study, the subject will return to their eye care professional for their routine eye care.

#### 11 ADVERSE EVENTS AND DEVICE DEFICIENCIES

#### 11.1 General Information

An AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the investigational medical device (test article). Refer to the Glossary of Terms and figures below for categories of AEs and SAEs.

Figure 11–1 Categorization of All AEs




Status: Effective 

Figure 11-2 Categorization of All SAE



#### SAEs

In addition to reporting all AEs (serious and non-serious) meeting the definitions, the Investigator must report any occurrence of the following as an SAE:

- An ocular infection including a presumed infectious ulcer with any of the following characteristics\*:
  - Central or paracentral location
  - Penetration of Bowman's membrane
  - o Infiltrates > 2 mm diameter
  - Iritis
  - o Increase in intraocular pressure
  - Culture positive for microorganisms
  - Increasing size or severity at subsequent visits
- Any central or paracentral corneal event (such as neovascularization) that results in permanent opacification
- Hypopyon


Status: Effective 

- Hyphema
- Neovascularization within the central 6 mm of the cornea
- Permanent vision loss as defined by loss of 2 or more lines of BCVA from enrollment visit (Visit 1) that fails to resolve
- Uveitis (anterior, intermediate, or posterior)
- Corneal abrasion affecting  $\geq 50\%$  of corneal surface area

\*NOTE: Culture samples (from the subject's eyes, lenses, etc) must be taken at Investigator's discretion [as described in the MOP; and documented in the narrative section(s) of the corresponding ADE-SAE eCRF] for any suspected ocular infection, including infiltrates with overlying epithelial defect.

#### Significant Non-Serious AE

A significant non-serious AE is a device-related, non-sight threatening AE that warrants discontinuation of any contact lens wear for greater than or equal to 2 weeks. In addition, the Investigator must report any occurrence of the following as a Significant Non-Serious Adverse Event:

- Peripheral non-progressive non-infectious ulcers
- All symptomatic corneal infiltrative events
- Corneal staining score greater than or equal to Grade 3 (Refer to MOP for grading scales)
- Temporary vision loss as defined by loss of 2 or more lines of BCVA from enrollment visit (Visit 1) that persists for 2 or more weeks
- Neovascularization score greater than or equal to Grade 2 (Refer to MOP for grading scales)

The above events are based upon the categories provided in ISO 11980 and the US FDA Premarket Notification (510(k)) Guidance Document for Daily Wear Contact Lenses.

#### **Device Deficiencies**

A device deficiency is inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety, or performance. A device deficiency may or may not be associated with subject harm (ie, ADE or SADE); however, not all ADEs or SADEs are due to a device deficiency. The Investigator should determine the applicable category listed in the


Status: Effective 

Device Deficiency eCRF for the identified or suspect device deficiency and report any subject harm separately. Examples of device deficiencies include the following:

- Failure to meet product specifications (eg, incorrect lens power/diameter/base curve/color)
- Lens cloudy
- Lens surface/edge defect
- Torn lens during handling/in pack
- Packaging deficit (eg, mislabeled product)
- Suspect product contamination
- Lack of performance

## 11.2 Monitoring for AEs

At each visit, after the subject has had the opportunity to spontaneously mention any problems, the Investigator should inquire about AEs by asking the standard questions:

- "Have you had any health problems since your last study visit?"
- "Have there been any changes in the medicines you take since your last study visit?"

Changes in *any protocol-specific parameters and/or questionnaires* evaluated during the study are to be reviewed by the Investigator. Any untoward (unfavorable and unintended) change in *a protocol-specific parameter or questionnaire response* that is clinically relevant, in the opinion of the Investigator, is to be reported as an AE. These clinically relevant changes will be reported regardless of causality.

# 11.3 Procedures for Recording and Reporting

AEs are collected from the time of informed consent. Any pre-existing medical conditions or signs/symptoms present in a subject prior to the start of the study (ie, before informed consent is signed) are not considered AEs in the study and should be recorded in the Medical History section of the eCRF.

In addition, temporary lens awareness or visual changes during the fitting process are not considered AEs if the Investigator assesses that the symptom(s) can reasonably resolve within the anticipated adaptation period.

For each recorded event, the ADEs and SAEs documentation must include: date of occurrence, severity, treatment (if applicable), outcome, and assessments of the seriousness


Status: Effective 

and causality. In addition, the Investigator must document all device deficiencies reported or observed with test and control products on the Device Deficiency eCRF. The site must submit all available information on ADEs, SAEs, and device deficiencies to the Study Sponsor immediately as follows:

- ADEs or SAEs are documented on the *Serious Adverse Event and Adverse Device Effect* eCRF within 24 hours of the Investigator's or site's awareness.
- Device deficiencies are documented on the *Device Deficiency* eCRF within 24 hours of the Investigator's or site's awareness.
- A printed copy of the completed *Serious Adverse Event and Adverse Device Effect* and/or *Device Deficiency* eCRF must be included with product returns.
- Additional relevant information after initial reporting must be entered into the eCRF as soon as the data become available.
- Document any changes to concomitant medications on the appropriate eCRFs.
- Document all relevant information from Discharge Summary, Autopsy Report,
   Certificate of Death, etc, if applicable, in narrative section of the Serious Adverse
   Event and Adverse Device Effect eCRF.

*Note:* Should the EDC system become non-operational, the site must complete the appropriate paper *Serious Adverse Event and Adverse Device Effect* and/or *Device Deficiency* Form. The completed form is emailed to the Study Sponsor at <a href="mass.safety@alcon.com">msus.safety@alcon.com</a> according to the timelines outlined above; however, the reported information must be entered into the EDC system once it becomes operational.

Additionally, any AEs and device deficiencies for non-study marketed products (ie, CLEAR CARE, be considered and processed as spontaneous (following the postmarket vigilance procedures) and should be communicated to the product's manufacturer as per local requirements.

Study Sponsor representatives may be contacted for any protocol related question; their contact information is provided in the MOP that accompanies this protocol.

Further, depending upon the nature of the AE or device deficiency being reported, the Study Sponsor may request copies of applicable portions of the subject's medical records. The Investigator must also report all AEs and device deficiencies that could have led to a SADE according to the requirements of regulatory authorities or IRB/IEC.


Status: Effective 

#### **Intensity and Causality Assessments**

Where appropriate, the Investigator must assess the intensity (severity) of the AE based upon medical judgment with consideration of any subjective symptom(s), as defined below:

#### Intensity (Severity)

Mild An AE is mild if the subject is aware of but can easily tolerate the sign or

symptom.

Moderate An AE is moderate if the sign or symptom results in discomfort significant

enough to cause interference with the subject's usual activities.

Severe An AE is severe if the sign or symptom is incapacitating and results in the

subject's inability to work or engage in their usual activities.

For every AE in the study, the Investigator must assess the causality (Related or Not Related to the medical device or study procedure). An assessment of causality will also be performed by Study Sponsor utilizing the same definitions, as shown below:

#### Causality

Related An AE classified as related may be either definitely related or possibly related

where a direct cause and effect relationship with the medical device or study procedure has not been demonstrated, but there is a reasonable possibility that

the AE was caused by the medical device or study procedure.

Not Related An AE classified as not related may either be definitely unrelated or simply

unlikely to be related (ie, there are other more likely causes for the AE).

The Study Sponsor will assess the AEs and may upgrade the Investigator's assessment of seriousness and/or causality. The Study Sponsor will notify the Investigator of any AEs that are upgraded from non-serious to serious or from unrelated to related.

Additionally, the Study Sponsor shall immediately conduct an evaluation of any unanticipated adverse device effect, including anticipated adverse events that occur in unanticipated severity or frequency. The results of this evaluation will be reported to the FDA, the IRB, and participating Investigators within 10 working days upon receiving notification of the effect.


Status: Effective 

## 11.4 Return Product Analysis

Investigational product associated with device deficiencies and/or product related AEs (ie, ADE or SADE) will be returned for investigation as detailed in the MOP.

## 11.5 Unmasking of the Study Treatment

Masked information on the identity of the assigned medical device should not be disclosed during the study. If the treatment code needs to be broken in the interest of subject safety, the Investigator is encouraged to contact an appropriate Study Sponsor representative prior to unmasking the information if there is sufficient time. Dependent upon the individual circumstances (ie, medical emergency), the code may be broken prior to contact with the Study Sponsor. The Study Sponsor must be informed of all cases in which the code was broken and of the circumstances involved. Additionally, the Study Sponsor may be required to unmask the information in order to fulfill expedited regulatory requirements.

## 11.6 Follow-Up of Subjects with AEs

The Investigator is responsible for adequate and safe medical care of subjects during the study and for ensuring that appropriate medical care and relevant follow-up procedures are maintained after the study.

The Investigator should provide the Study Sponsor with any new safety information (which includes new AEs and changes to previously reported AEs) that may affect the safety evaluation of the device. For AEs that are unresolved/ongoing at time of subject exit from study, any additional information received at follow-up should be documented in the eCRFs up to study completion (ie, database lock).

Any additional data received up to 3 months after subject discontinuation or exit must be documented and available upon the Study Sponsor's request. All complaints received after this time period will be considered and processed as spontaneous (following the postmarket vigilance procedures) and should be communicated to the medical device's manufacturer as per local requirements, as applicable.

The Investigator should also report complaints on non-Alcon products directly to the manufacturer as per the manufacturer's instructions or local regulatory requirements.

# 11.7 Pregnancy in the Clinical Study

Women of childbearing potential or women who are pregnant at the time of study entry are not excluded from participation. Pregnancy should be included in the Medical History section


Status: Effective 

of the eCRF when a pregnant woman enters the study or if a woman becomes pregnant during the study. Pregnancy is not reportable as an AE; however, complications may be reportable and will be decided on a case-by-case basis.

#### 12 ANALYSIS PLAN

Any deviations to the analysis plan will be updated during the course of the study as part of a protocol amendment or will be detailed in the clinical study report.

All analyses will be conducted according to the applicable statistical analysis plan.

## 12.1 Subject Evaluability

Final subject evaluability must be determined prior to breaking the code for masked treatment assignment and locking the database, based upon the Deviations and Evaluability Plan.

## 12.2 Analysis Sets

Five analysis sets will be defined:

- a) All Enrolled all subjects signing the informed consent form
- b) Enrolled Dispensed subjects/eyes from All Enrolled that have been exposed to study lenses (not considering trial-fit lenses prior to randomization)
- c) Enrolled Not Dispensed subjects/eyes from All Enrolled that have not been exposed to study lenses (not considering trial-fit lenses prior to randomization)
- d) Completed Enrolled Dispensed subjects/eyes completing the study
- e) Discontinued Enrolled Dispensed subjects/eyes not complete the study

# 12.3 Demographic and Baseline Characteristics

Demographic information, recent lens-wearing experience (including wear modality and wear success), and habitual lens information will be presented by lens group and overall for the All Enrolled analysis set.

Baseline data will be summarized by lens group, for Completed and Discontinued analysis sets separately, as applicable.


Status: Effective 

## 12.4 Effectiveness Analyses

For each of the primary and supportive effectiveness endpoints, separate summary tables will be prepared, when applicable, for the Completed and the Discontinued analysis sets as follows:

- Completed Control (eyes/subjects)
- Completed Test (eyes/subjects)
- Discontinued Control (eyes/subjects)
- Discontinued Test (eyes/subjects)

No inferential testing will be performed on effectiveness endpoints, and format of the reporting tables will follow FDA's 510(k) guidance document (Clinical Appendix C, Summary of Reporting Tables) as well as the ISO guidance as specified in Section A.3 (Reporting of results) of ISO 11980:2012.

## 12.4.1 Analysis of Primary Effectiveness Endpoint(s)

The primary objective of this study is to evaluate visual acuity of the investigational soft contact lens compared to the commercially available Biofinity soft contact lens.

The primary effectiveness endpoint is distance VA with study lenses, collected in Snellen, for each eye. Conversion will be made to the logMAR scale.

# **12.4.1.1** Statistical Hypotheses

No hypothesis testing of the primary effectiveness endpoint is planned.




Effective Date: 08-Nov-2019

# 12.4.2.1 Statistical Hypotheses and Model

Alcon - Business Use Only Protocol - Clinical

No hypothesis testing of the supportive effectiveness endpoints is planned.

# 12.4.2.2 Analysis Methods

For each of the supportive effectiveness endpoints, descriptive summary statistics will be computed according to the scale of measurement.

# 12.5 Handling of Missing Data

All data obtained in evaluable subjects/eyes will be used. No imputation for missing values will be carried out.

Incidence and reasons for discontinuation by lens group will be tabulated at each visit and overall.


Status: Effective 

## 12.6 Safety Analyses

The safety endpoints are:

- AEs
- Biomicroscopy findings
- Device deficiencies

There are no safety hypotheses planned in this study. The focus of the safety analysis will be a comprehensive descriptive assessment of occurrence of AE as well as the other listed parameters.

Descriptive summaries (counts and percentages) for ocular and nonocular AEs will be presented by Medical Dictionary for Regulatory Activities Preferred Terms, for Completed and Discontinued sets. A listing containing details of the AEs will also be provided. Each biomicroscopy parameter will be tabulated by its grade, on Completed and Discontinued analysis sets. Frequency for each device deficiency category will be presented and a supporting listing will be provided.

## 12.7 Interim Analyses and Reporting

There are no plans to conduct an interim analysis.

# 12.8 Sample Size Justification

Sample size is based upon the following:

- Premarket Notification (510(k)) Guidance Document for Daily Wear Contact Lenses –
  at least 50 evaluable subjects to be followed for at least 3 months, for claim of
  substantial equivalence for a lens with different repeating monomer Units (new Parent
  USAN). In addition, a 2:1 ratio in Test vs Control evaluable subject allocation should
  be adopted.
- ISO 11980:2012 50 completed subjects in Test, for 3 months. Either 2:1 or 1:1 ratio of Test to Control can be accepted.

# 13 DATA HANDLING AND ADMINISTRATIVE REQUIREMENTS

# 13.1 Subject Confidentiality

The Investigator must ensure that the subject's anonymity is maintained throughout the course of the study. In particular, the Investigator must keep an enrollment log with


Status: Effective 

confidential identifying information that corresponds to the subject numbers and initials of each study participant. At the end of the clinical study, the Study Sponsor will collect a copy of the enrollment log *without any identifying subject information*. All documents submitted to the Study Sponsor will identify the subjects exclusively by number and demographic information. No other personally identifying information will be transmitted to the Study Sponsor.

The Study Sponsor may release anonymized study data to external researchers for purposes of future research directly related to the study objectives, or future research that is beyond the scope of the current study objectives. The Informed Consent Form explains this to study subjects. Anonymization means that all identifiable information will be removed from the dataset and all links to the subjects in the study will be removed. Anonymization of the data will maintain confidentiality of the subjects who participate in the study so that they cannot be identified by external researchers. The anonymized data set will contain records from all of the subjects in the current study, but the anonymization process might change the data set in some ways, so external researchers will be informed that they might not be able to duplicate some of the results from this study.

## 13.2 Completion of Source Documents and Case Report Forms

The nature and location of all source documents will be identified to ensure that original data required to complete the CRFs exist and are accessible for verification by the site monitor, and all discrepancies shall be appropriately documented via the query resolution process. Site monitors are appointed by the Study Sponsor and are independent of study site staff.

If electronic records are maintained, the method of verification must be determined in advance of starting the study.

At a minimum, source documents include the following information for each subject:

- Subject identification (name, sex, race/ethnicity)
- Documentation of subject eligibility
- Date of informed consent
- Dates of visits
- Documentation that protocol specific procedures were performed
- Results of study parameters, as required by the protocol
- IP accountability records


Status: Effective 

- Documentation of AEs and other safety parameters (if applicable)
- Records regarding medical histories and the use of concomitant therapies prior to and during the study
- Date of study completion and reason for early discontinuation, if applicable

It is required that the author of an entry in the source documents be identifiable. Direct access to source documentation (medical records) must be allowed for the purpose of verifying that the data recorded on the CRF are consistent with the original source data.

Only designated individuals at the site will complete the CRFs. The CRFs must be completed at regular intervals following the clinical study visit schedule. It is expected that all data reported have corresponding entries in the source documents. The Principal Investigator is responsible for reviewing and certifying that the CRFs are accurate and complete. The only subject identifiers recorded on the CRFs will be subject number and subject demographic information.

#### 13.3 Data Review and Clarifications

A review of CRF data to the subject's source data will be completed by the site monitor to ensure completeness and accuracy. After the CRFs have been completed, additional data clarifications and/or additions may be needed as a result of the data cleaning process. Data clarifications are documented and are part of each subject's CRF.

# 13.4 Sponsor and Monitoring Responsibilities

The Study Sponsor will designate a monitor to conduct the appropriate site visits at the appropriate intervals according to the study monitoring plan. The clinical investigation will be monitored to ensure that the rights and well-being of the subjects are protected, the reported data are accurate, complete, and verifiable from the source documents, and the study is conducted in compliance with the current approved protocol (and amendments[s], if applicable), with current GCP, and with applicable regulatory requirements.

The site may not screen subjects or perform the informed consent process on any subject until it receives a notification from an appropriate Study Sponsor representative that the site may commence conducting study activities. Monitoring will be conducted periodically while the clinical study is ongoing. Monitoring methods may include site visits, telephone, written, and fax correspondence. Close-out visits will take place after the last visit of the last subject at the site.


Status: Effective 

A Coordinating Investigator may be identified by the Study Sponsor to review and endorse the final study report. In cases where a Coordinating Investigator is engaged, the Study Sponsor will select the Coordinating Investigator based upon their experience, qualifications, active study participation, and their willingness and availability to take on this role.

#### 13.5 Regulatory Documentation and Records Retention

The Investigator is required to maintain up-to-date, complete regulatory documentation as indicated by the Study Sponsor and the Investigator's files will be reviewed as part of the ongoing study monitoring. Financial information is to be kept separately.

Additionally, the Investigator must keep study records and source documents consistent with the terms of the clinical study agreement with the Study Sponsor. If the Investigator retires, relocates, or for any other reason withdraws from responsibility of keeping the study records, then the Study Sponsor must be notified and suitable arrangements made for retention of study records and source documents needed to comply with national and international regulations.

## 13.6 Quality Assurance and Quality Control

The Study Sponsor will secure agreement from all involved parties to ensure direct access to all study-related sites, source data and documents, and reports for the purpose of monitoring and auditing by the Study Sponsor, and inspection by domestic and foreign regulatory authorities. Quality control will be applied to each stage of data handling to ensure that all data are reliable and have been processed correctly. Agreements made by the Study Sponsor with the Investigator/Institution and any other parties involved in the clinical study will be provided in writing as part of the protocol or as a separate agreement.

#### 14 ETHICS

This clinical study must be conducted in accordance with the ethical principles contained within:

- The Declaration of Helsinki, and in compliance with the ICH E6 GCP Consolidated Guideline, ISO 14155:2011, and the applicable US FDA 21 CFR Regulations.
- SOPs of the Study Sponsor and contract research organizations participating in the conduct of the clinical study and all other applicable regulations.
- Notifications and timelines for reporting protocol deviations should be based upon applicable Ethics Committee requirements.


Status: Effective 

The Investigator must ensure that all personnel involved in the conduct of the study are qualified to perform their assigned responsibilities through relevant education, training, and experience. The Investigator and all clinical study staff must conduct the clinical study in compliance with the protocol. Deviations from this protocol, regulatory requirements, and/or GCP must be recorded and reported to the Sponsor prior to database lock. If needed, corrective and preventive action should be identified, implemented, and documented within the study records. Use of waivers to deviate from the clinical protocol is prohibited.

Before clinical study initiation, this protocol, the informed consent form, any other written information given to subjects, and any advertisements planned for subject recruitment must be approved by an IRB/IEC. The Investigator must provide documentation of the IRB/IEC approval to the Study Sponsor. The approval must be dated and must identify the applicable protocol, amendments (if any), informed consent form, assent form (if any), all applicable recruiting materials, written information for subject, and subject compensation programs. The IRB/IEC must be provided with a copy of the IB, any periodic safety updates, and all other information as required by local regulation and/or the IRB/IEC. At the end of the study, the Investigator must notify the IRB/IEC about the study's completion. The IRB/IEC also must be notified if the study is terminated prematurely. Finally, the Investigator must report to the IRB/IEC on the progress of the study at intervals stipulated by the IRB/IEC.

Voluntary informed consent must be obtained in writing from every subject and the process shall be documented before any procedure specific to the clinical investigation is applied to the subject. The Investigator must have a defined process for obtaining consent. Specifically, the Investigator, or their delegate, must explain the clinical study to each potential subject and the subject must indicate voluntary consent by signing and dating the approved informed consent form. The subject must be provided an opportunity to ask questions of the Investigator, and if required by local regulation, other qualified personnel. The Investigator must provide the subject with a copy of the consent form written in a language the subject understands. The consent document must meet all applicable local laws and provide subjects with information regarding the purpose, procedures, requirements, and restrictions of the study, along with any known risks and potential benefits associated with the IP and the study, the available compensation, and the established provisions for maintaining confidentiality of personal, protected health information. Subjects will be told about the voluntary nature of participation in the study and must be provided with contact information for the appropriate individuals should questions or concerns arise during the study. The subject also must be told that their records may be accessed by appropriate authorities and Sponsor-designated personnel. The Investigator must keep the original, signed copy of the consent (file in


Status: Effective 

subject's medical records) and must provide a duplicate copy to each subject according to local regulations.

The Study Sponsor assures that the key design elements of this protocol will be registered on www.clinicaltrials.gov as required by current regulations and, if applicable, other public databases as required by local country regulations. In addition, results of this study will be made publicly available on www.clinicaltrials.gov regardless of outcome as required by current regulations and, if applicable, in other public databases as required by local country regulations.

#### 15 REFERENCES

## 15.1 References Applicable for All Clinical Studies

- ISO 11980:2012 Ophthalmic optics Contact lenses and contact lens care products -Guidance for clinical investigations
- ISO 14155:2011 Clinical investigation of medical devices for human subjects Good clinical practice

## 15.1.1 US References Applicable for Clinical Studies

- 21 CFR Part 11 Electronic Records; Electronic Signatures
- 21 CFR Part 50 Protection of Human Subjects
- 21 CFR Part 56 Institutional Review Boards
- 21 CFR Part 812 Investigational Device Exemptions
- 21 CFR Part 54 Financial Disclosure by Clinical Investigators
- The California Bill of Rights

# 15.2 Additional References for This Clinical Study

 Premarket Notification [510((k)] Guidance Document for Daily Wear Contact Lenses, May 1994


Status: Effective